CLINICAL TRIAL: NCT06516354
Title: Evaluation of Obstructive Sleep Apnea (OSA) Using Portable Sleep Testing (PST) Devices on an Inpatient Stroke Unit
Acronym: OSA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment; no patients were enrolled
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AHC6601
Record Dates: First submitted 2018-02-21; First posted 2024-07-23 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Portable Sleep Apnea Screening (Other): Application of portable sleep apnea screening device on inpatient stroke/TIA patients for at least 5 hours of sleep in one night or 8 hours of sleep over 2 consecutive nights.
  Interventions: Device: Portable sleep apnea screening

INTERVENTIONS:
Device: Portable sleep apnea screening — Screening of stroke and TIA patients on the stroke inpatient unit using theSTOP BANG questionnaire and portable sleep testing (PST) during inpatient hospitalization, early interpretation of PST results by neurology with prescribed treatment upon discharge from hospital

SUMMARY:
The purpose of this study is to evaluate the feasibility of testing patients for OSA within the inpatient setting. As part of this program, the investigators are proposing early access to a sleep apnea treatment plan, potentially lowering the risk for future stroke symptoms, and preventing lost to follow up of patients for treatment since sleep disordered breathing is primarily considered a disorder that is managed in an outpatient setting.

Hypothesis: Early identification of sleep apnea as a modifiable stroke risk factor (SRF) for acute ischemic stroke (AIS) and transient ischemic attack (TIA) patients using the STOP BANG questionnaire and portable sleep testing (PST) during inpatient hospitalization, will allow early identification of patients at risk for sleep disordered breathing, early diagnosis of sleep apnea, and earlier prescribed treatment prior to discharge.

DETAILED DESCRIPTION:
Currently the standard of care at Lutheran General Hospital for patients does not include a STOP BANG pre-screening assessment, and portable sleep testing (PST) to identify sleep disordered breathing as a risk factor for AIS and TIA. Initially, patients will be asked questions if they have a history of OSA diagnosis, and if ever have been treated with a form of PAP. If the response is no, then the patient will be prescreened using the STOP BANG assessment tool and review of eligibility requirements. If positive STOP BANG and patient meets eligibility, the patient will have the PST device registered and the Watermark ARES 610 will be applied by the sub investigators. The patient will then undergo a portable sleep study which measures nasal pressure, respiratory effort, oxygen saturation, electrocardiogram and body position. If the device needs adjustment during sleep it can be adjusted by patient or Nursing Care Technician. The next morning the PST device, which is removed by sub investigators, will be delivered to the Sleep Laboratory, downloaded by the sleep technician in Sleep Lab, and data transmitted via the hospital network to the sleep specialist (Primary Investigator) for interpretation. If the PST study is interpreted as positive this will initiate a treatment plan by the sleep specialist for prescription of PAP and/or follow up. This patient who is positive will not require an additional polysomnogram for confirmation of the sleep apnea in the outpatient setting. If the result is inconclusive, but highly suspicious, this may require additional outpatient testing.

ELIGIBILITY:
Inclusion Criteria:

* • Acute ischemic stroke (AIS) or transient ischemic attack (TIA) diagnosis during hospitalization

  * Patient on neurology stroke care unit (10 Tower)
  * Consenting adults (≥ 18 years old)

    o For subjects unable to effectively communicate or sign consent due to stroke symptoms, informed consent will be obtained from LAR (legally authorized representative)
  * Positive STOP BANG screen
  * NIHSS 0-25 (higher NIHSS scores may require application of the PST other than by the patient)

Exclusion Criteria:

* • Patients who receive sedation within 24 hours of portable sleep testing

  * Refusal to sign informed consent
  * Non English speaking patient
  * Inability to designate Legally Authorized Representative (LAR) for consent
  * Participation in other ongoing neurothrombectomy research studies
  * Time from symptom onset to emergency department arrival ˃ 72 hours
  * Respiratory distress requiring mechanical ventilation or supplemental oxygen at the time of pre screening
  * Cardiac or respiratory arrest within past 3 months
  * Myocardial infarction (MI) within the past 3 months
  * Any unstable medical condition likely to interfere with participation of portable sleep testing
  * Life expectancy less than 6 months
  * Prior known diagnosis of OSA
  * Currently treated with CPAP device
  * Pregnant and breastfeeding women
  * Prisoners
* Patients unable to complete at least 5 hours of sleep per one night or 8 hours of sleep over 2 nights

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-28 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
STOP BANG tool | 90 days
  Positive screening on STOP BANG tool for sleep disordered breathing completed during inpatient hospitalization prior to discharge.
Portable Sleep Testing | 90 days
  Positive screening on Portable Sleep Testing (PST) for sleep disordered breathing completed during inpatient hospitalization prior to discharge.

SECONDARY OUTCOMES:
Follow up compliance | 120 days
  Phone call with patient to assess compliance and tolerability to treatment plan
Follow up readmission rate | 120 days
  Hospital readmission due to stroke from the Crimson database

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Tumashova, MD, Principal Investigator — Advocate Medical Group Neurologist
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chernyshev OY, McCarty DE, Moul DE, Liendo C, Caldito GC, Munjampalli SK, Kelley RE, Chesson AL Jr. A pilot study: portable out-of-center sleep testing as an early sleep apnea screening tool in acute ischemic stroke. Nat Sci Sleep. 2015 Oct 20;7:127-38. doi: 10.2147/NSS.S85780. eCollection 2015. PMID 26527904
- [Background] Davis AP, Billings ME, Longstreth WT Jr, Khot SP. Early diagnosis and treatment of obstructive sleep apnea after stroke: Are we neglecting a modifiable stroke risk factor? Neurol Clin Pract. 2013 Jun;3(3):192-201. doi: 10.1212/CPJ.0b013e318296f274. PMID 23914326
- [Background] Goldstein LB, Bushnell CD, Adams RJ, Appel LJ, Braun LT, Chaturvedi S, Creager MA, Culebras A, Eckel RH, Hart RG, Hinchey JA, Howard VJ, Jauch EC, Levine SR, Meschia JF, Moore WS, Nixon JV, Pearson TA; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Epidemiology and Prevention; Council for High Blood Pressure Research,; Council on Peripheral Vascular Disease, and Interdisciplinary Council on Quality of Care and Outcomes Research. Guidelines for the primary prevention of stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2011 Feb;42(2):517-84. doi: 10.1161/STR.0b013e3181fcb238. Epub 2010 Dec 2. PMID 21127304
- [Background] Johnson KG, Johnson DC. Frequency of sleep apnea in stroke and TIA patients: a meta-analysis. J Clin Sleep Med. 2010 Apr 15;6(2):131-7. PMID 20411688
- [Background] Kauta SR, Keenan BT, Goldberg L, Schwab RJ. Diagnosis and treatment of sleep disordered breathing in hospitalized cardiac patients: a reduction in 30-day hospital readmission rates. J Clin Sleep Med. 2014 Oct 15;10(10):1051-9. doi: 10.5664/jcsm.4096. PMID 25317084
- [Background] King S, Cuellar N. Obstructive Sleep Apnea as an Independent Stroke Risk Factor: A Review of the Evidence, Stroke Prevention Guidelines, and Implications for Neuroscience Nursing Practice. J Neurosci Nurs. 2016 Jun;48(3):133-42. doi: 10.1097/JNN.0000000000000196. PMID 27136407
- [Background] Redline S, Yenokyan G, Gottlieb DJ, Shahar E, O'Connor GT, Resnick HE, Diener-West M, Sanders MH, Wolf PA, Geraghty EM, Ali T, Lebowitz M, Punjabi NM. Obstructive sleep apnea-hypopnea and incident stroke: the sleep heart health study. Am J Respir Crit Care Med. 2010 Jul 15;182(2):269-77. doi: 10.1164/rccm.200911-1746OC. Epub 2010 Mar 25. PMID 20339144
- [Result] Aparicio, HJ. Stroke Unit Evaluation of Sleep Apnea: Validating Screening Tools and the Use of a Portable Sleep Study Device. 2016 International Stroke Conference, Los Angeles, CA 17 Feb 2016 Presentation